CLINICAL TRIAL: NCT06525675
Title: Study to Evaluate the Extended Overall Survival From PARSIFAL Trial: Efficacy and Safety of Palbociclib in Combination With Fulvestrant or Letrozole in Patient With HER2-/ER+ Metastatic Breast Cancer (The PARSIFAL-LONG Study)
Brief Title: Study to Evaluate the Extended Overall Survival (OS) Data From PARSIFAL Study (The PARSIFAL-LONG Study)
Status: Completed | Type: Observational
Sponsor: MedSIR (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: MEDOPP507
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer; Luminal Breast Cancer; HER2-negative Breast Cancer; ER-positive Breast Cancer
Keywords: breast cancer; metastatic breast cancer; luminal breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Letrozole; palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fulvestrant plus palbociclib (interventional arm): Postmenopausal women and premenopausal women receiving Luteinizing Hormone-Releasing Hormone (LHRH) analogues, aged ≥ 18 years with ER positive and HER2 negative locally advanced or metastatic breast cancer that had not received any therapy for the metastatic disease. Patients are not eligible if they are candidates for a local treatment with a radical intention. Subjects must have histologic confirmation of the estrogen and/or progesterone-positive and HER2 negative receptors breast cancer. Evidence of measurable or evaluable metastatic disease is required.
  Interventions: Drug: Fulvestrant Injectable Product; Drug: Palbociclib 125mg
- Letrozole plus palbociclib (control arm): Postmenopausal women and premenopausal women receiving Luteinizing Hormone-Releasing Hormone (LHRH) analogues, aged ≥ 18 years with ER positive and HER2 negative locally advanced or metastatic breast cancer that had not received any therapy for the metastatic disease. Patients are not eligible if they are candidates for a local treatment with a radical intention. Subjects must have histologic confirmation of the estrogen and/or progesterone-positive and HER2 negative receptors breast cancer. Evidence of measurable or evaluable metastatic disease is required.
  Interventions: Drug: Letrozole 2.5mg; Drug: Palbociclib 125mg

INTERVENTIONS:
Drug: Fulvestrant Injectable Product — 500 mg fulvestrant on days 1, 14, 28, and once monthly thereafter, administered intramuscularly.
  Other Names: Faslodex®
  Groups: Fulvestrant plus palbociclib (interventional arm)
Drug: Letrozole 2.5mg — 2.5 mg letrozole per day, administered orally (continuous treatment)
  Other Names: Letrozole
  Groups: Letrozole plus palbociclib (control arm)
Drug: Palbociclib 125mg — orally administration 125 mg palbociclib per day (in cycles of 3 weeks of treatment followed by 1 week off)
  Other Names: PD-0332991

SUMMARY:
The goal of this study is to evaluate the extended Overall Survival (OS) from PARSIFAL trial - NCT02491983 focused on the efficacy and safety of palbociclib in combination with fulvestrant or letrozole in patients with Human Epidermal growth factor Receptor 2 (HER2)-negative, Endocrine Receptor (ER)-positive metastatic breast cancer. It was designed to test the superiority of fulvestrant plus palbociclib compared with letrozole plus palbociclib first and then the non-inferiority of fulvestrant plus palbociclib compared with letrozole plus palbociclib if the superiority objective was not achieved.

DETAILED DESCRIPTION:
This is an observational, international multi-center study with the objective to evaluate the extended overall survival from PARSIFAL trial (NCT02491983) analyzing the efficacy and safety of palbociclib in combination with fulvestrant or letrozole in patients with HER2-negative, ER-positive locally advanced or metastatic breast cancer. The patients included in this trial were previously randomized in PARSIFAL trial and did not withdraw consent to participate in the PARSIFAL clinical trial. The primary objective is to compare the efficacy (in terms of OS) of palbociclib in combination with fulvestrant (interventional arm) versus palbociclib plus letrozole (control arm) during extended follow-up of PARSIFAL trial and the secondary objectives are to assess the extended efficacy, of palbociclib combined with fulvestrant or letrozole in terms of progression-free survival (PFS), to estimate the extended efficacy, of palbociclib combined with endocrine therapy (fulvestrant or letrozole) in terms of OS and PFS and to assess the subsequent antineoplastic therapies to palbociclib combined with fulvestrant or letrozole in this population. The PARSIFAL-LONG study is non-interventional. There are no protocol-mandated visits or procedures associated with the study. In this study the data required to document the defined study endpoints will be collected using the medical histories of patients accrued in the PARSIFAL study as data source. This additional data will be analyzed along with the database of PARSIFAL trial. The estimated study duration is 24 months and the expected period for data validation, analysis, and reporting is around 4 more months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously randomized in the PARSIFAL trial (N = 486).
2. Patients did not withdraw consent to participate in the PARSIFAL clinical trial.

Patients randomized in PARSIFAL trial had to meet the following inclusion criteria:

1. Postmenopausal women, as defined by any of the following criteria:

   * Age 60 or over
   * Age 45 to 59 years and meets ≥1 of the following criteria: amenorrhea for ≥ 24 months or amenorrhea for < 24 months and follicle-stimulating hormone within the postmenopausal range (including patients with hysterectomy, prior hormone replacement therapy or chemotherapy-induced amenorrhea).
   * Over 18 years of age and bilateral oophorectomy

   OR:

   Premenopausal women provided they are being treated with LHRH analogues for at least 28 days prior to study entry.
2. Eastern Cooperative Oncology Group (ECOG) score lower or equal to 2.
3. Histologically confirmed recurrent ER-positive (oestrogen and/or progesterone) HER2-negative locally advanced or metastatic BC patients (Breast cancer that have at least 1% of cells staging positive for ER should be considered ER-positive according to National Comprehensive Cancer Network (NCCN) and American Society of Clinical Oncology (ASCO) guidelines.
4. Patients should not be candidates for a local treatment with a radical intention.
5. No prior hormonal or chemotherapy line in the metastatic setting.
6. Patient must have measurable (according to RECIST 1.1) or non-measurable disease with these exceptions:

   1. Patients with only blastic bone lesions are not eligible.
   2. Patients with only pleural, peritoneal, or cardiac effusion, or meningeal carcinomatosis are not eligible.
7. Life expectancy grater or equal to 12 weeks.
8. Adequate organ function:

   1. Hematological: White blood cell (WBC) count >3.0 x 109/L, absolute neutrophil count (ANC) >1.5 x 109/L, platelet count >75.0 x109/L, and hemoglobin >10.0 g/dL (>6.2 mmol/L)
   2. Hepatic: bilirubin < 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (ALP), aspartate transaminase (AST), and alanine transaminase (ALT) <2.5 times ULN. Patients with ALP ≥2.5 times ULN are eligible if ALP abnormalities are unequivocally related to bone lesions (radiological assessments performed within 4 weeks prior to randomization demonstrated bone metastatic disease).
   3. Renal: serum creatinine < 1.5 x ULN.
9. Exhibit patient compliance and geographic proximity that allow for adequate follow-up.
10. Patient has been informed about the nature of study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.
11. No other malignancies within the past five years except adequate treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
12. Resolution of all acute toxic effects of prior anti- cancer therapy or surgical procedures to NCI- CTCAE version 4.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
13. Patient has been informed about the translational sub-study and has agreed to participate in the collection of blood and tumor tissue samples by signing the Informed Consent form.

Exclusion Criteria:

Patients were excluded from the PARSIFAL trial if they met any of the following criteria:

1. ER or HER2 unknown disease.
2. HER2-positive disease based on local laboratory results (performed by immunohistochemistry/FISH)
3. Locally advanced breast cancer candidate for a radical treatment.
4. Prior endocrine therapy in the metastatic setting. (Neo)/Adjuvant endocrine therapy is allowed only if the disease-free interval between the end of endocrine therapy and the appearance of metastases in higher than 12 months.
5. Patients with rapidly progressive visceral disease or visceral crisis.
6. Have had a major surgery (defined as requiring general anesthesia) or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the study.
7. Patients with an active, bleeding diathesis.
8. Have a serious concomitant systemic disorder (e.g. active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator), previous history of bleeding diathesis, or anti-coagulation treatment (The use of low molecular weight heparin is allowed as long as it is used as prophylaxis).
9. Are unable to swallow tablets.
10. History of malabsorption syndrome or other condition that would interfere with enteral absorption.
11. Chronic daily treatment with corticosteroids with a dose of ≥ 10mg/day methylprednisolone equivalent (excluding inhaled steroids).
12. Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral oedema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (e.g., radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
13. Known hypersensitivity to letrozole, fulvestrant or any of their excipients, or to any palbociclib excipients.
14. Corrected QT Interval (QTc) >480 msec on basal assessments, personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
15. Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible women were aged 18 y or older with menopausal status and HER2-negative/ER-positive, unresectable, locally advanced, or metastatic breast cancer not treatable with curative intent. Patients had not received systemic therapy for advanced disease and had measurable or non measurable disease as defined by RECIST version 1.1. Endocrine therapy in the neoadjuvant or adjuvant setting was permitted if the patient had a disease-free interval of more than 12m from the completion of endocrine therapy. An Eastern Cooperative Oncology Group (ECOG) score of 0 to 2 and adequate organ function were also required. Key exclusion criteria were visceral crisis and prior treatment with a CDK4/6 inhibitor.
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 24 months
  Overall Survival (OS) is defined as the time from randomization until death from any cause in the palbociclib plus fulvestrant group versus the palbociclib plus letrozole group

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  Progression Free Survival (PFS) is defined as the time from randomization until objective tumor progression or death, as assessed by the investigator per RECIST v1.1, in the palbociclib plus fulvestrant group versus the palbociclib plus letrozole group
Overall Survival (OS) | 24 months
  Overall Survival (OS) is defined as the time from randomization until death from any cause, in the palbociclib plus endocrine therapy (fulvestrant or letrozole) treated patients
Progression Free Survival (PFS) | 24 months
  Progression Free Survival (PFS) is defined as the time from randomization until objective tumor progression or death, as assessed by the investigator per RECIST v1.1, in the palbociclib plus endocrine therapy (fulvestrant or letrozole) treated patients
Number of patients with the same subsequent antineoplastic therapy | 24 months
  Number of patients with the same subsequent antineoplasic therapy is described as the number of patients with the same antineoplastic therapy administered after the end of the treatment with palbociclib combined with endocrine therapy (fulvestrant or letrozole).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, Principal Investigator — Arnau de Vilanova Hospital
Locations (36):
- Czechia (2):
  - Onkologická klinika Fakultní nemocnice Olomouc, Olomouc
  - General University Hospital in Prague, Prague
- France (5):
  - Hopital Tenon, Paris
  - Hospital Europeo Georges Pompidou AP-HP, Paris
  - Institut Curie, Paris
  - Centre Paul Strauss, Strasbourg
  - Institut Universitaire du Cancer Toulouse, Toulouse, Toulouse
- Klinikum Dessau (MVZ) - Frauenheilkunde, Dessau, Germany
- Italy (4):
  - Istituti Ospitalieri Cremona, Cremona
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milano., Milan
  - Instituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo, Monza
- Spain (19):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital San Joan de Reus, Reus, Tarragona
  - Hospital Del Mar, Barcelona
  - Hospital Universitary Vall D´Hebron, Barcelona
  - Institut Català d' Oncologia L'Hospitalet (ICO), Barcelona
  - Institut Oncologic Baselga-Hospital Quiron Salud Barcelona, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Provincial de Castellón, Castellon
  - Hospital San Pedro Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - ICO Girona, Girona
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario La Paz, Madrid
  - CHUS Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Fundación Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Barts Cancer Institute, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Abertawe Bro Morgannwg University Local Health Board, Singleton Hospital, Swansea
  - Royal Cornwall Hospital NHS Trust, Truro